CLINICAL TRIAL: NCT01429376
Title: 1) Pulmonary Function in CHF; 2) COPD Prevalence, Underdiagnosis and Overdiagnosis in CHF Patients and Its Independent Predictors; 3) Are There Signs of Systemic Inflammation in CHF With or Without COPD?
Brief Title: Pulmonary Function, Chronic Obstructive Pulmonary Disease (COPD) Prevalence, and Systemic Inflammation in Chronic Heart Failure With or Without COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LTC-607-070409
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Heart Failure; Pulmonary Disease, Chronic Obstructive; Inflammation
Keywords: Chronic heart failure; Pulmonary function abnormalities/impairment; Restriction; Airway obstruction; Diffusion impairment; Pulmonary function tests; Chronic obstructive pulmonary disease (COPD); Prevalence; Overdiagnosis; Underdiagnosis; Systemic inflammation; Diagnostic Errors
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Inflammation; Airway Obstruction | interventions — Respiratory Physiological Phenomena; Hematologic Tests; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pulmonary function tests — Patients underwent several pulmonary function tests (spirometry, diffusion measurement, body plethysmography) according to the study protocol 1 month after the first blood sample. COPD was diagnosed post-bronchodilation according to GOLD guidelines. Patients with newly diagnosed COPD received standard treatment for COPD. Spirometry was repeated after 3 months of standard treatment for COPD in patients with newly diagnosed COPD to confirm persistent airway obstruction (COPD) and thus exclude asthma.
Other: Blood tests — First blood sample (day 1): NT-pro-BNP, sodium, potassium, urea, creatinin, glomerular filtration rate (GFR).
  Second blood sample (after 1 month): NT-pro-BNP, sodium, potassium, urea, creatinin, GFR, haemoglobin, and arterial blood gas analysis in patients with GOLD III COPD. For systemic inflammation substudy also high sensitivity CRP, leukocytes, and platelets.
  Third blood sample (after 3 months from second blood sample): NT-pro-BNP, sodium, potassium, urea, creatinin, and GFR.
Other: Questionnaires — Minnesota Living with Heart Failure Questionnaire (MLHFQ), modified Medical Research Council (MRC) dyspnoea scale, 10-point Borg dyspnoea score.
  All questionnaires were completed on the day of initial pulmonary function tests and three months later.
Other: Chest radiograph — Standard posteroanterior and lateral chest radiographs were performed and evaluated on the presence or absence of congestion and other conditions that belonged to the exclusion criteria.

SUMMARY:
The aim of the present study is:

1. To investigate pulmonary function abnormalities (restriction, obstruction, diffusion impairment, mixed pulmonary defects) in patients with chronic heart failure (CHF) and to determine which of these pulmonary abnormalities prevail and to what extent.
2. To determine the prevalence, underdiagnosis, and overdiagnosis of chronic obstructive pulmonary disease (COPD) as determined by spirometry and according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria in patients with CHF.
3. To investigate the presence of systemic inflammation, as measured by inflammatory parameters (leukocytes, platelets, high sensitivity CRP), in CHF patients with or without COPD.

DETAILED DESCRIPTION:
1. The impact of chronic heart failure (CHF) on pulmonary function is incompletely understood and remains controversial. It is difficult to separate the contribution of stable CHF from underlying pulmonary disease and other confounding influences, such as changes due to normal ageing, obesity, environmental exposure (mainly smoking), stability of disease, a history of coronary artery bypass grafting, and other conditions that can lead to pulmonary function abnormalities. Studies have shown that isolated or combined pulmonary function impairment, such as diffusion impairment, restriction, and to a much lesser extent airway obstruction are common in patients with CHF and can contribute to the perception of dyspnoea and exercise intolerance. Pulmonary dysfunction increases with the severity of heart failure and provides important prognostic information. Most investigators compared pulmonary function in CHF patients with normal predicted values or control subjects. However, there is only a small body of literature addressing the prevalence of different pulmonary function abnormalities in patients with CHF. In addition, these studies have included (potential) heart transplant recipients, who represent one extreme of the heart failure spectrum. The aim of the present study was to investigate the prevalence of pulmonary function abnormalities in patients with CHF and to determine which of these pulmonary abnormalities prevail and to what extent.
2. Chronic obstructive pulmonary disease (COPD) frequently coexists with CHF, leading to impaired prognosis as well as diagnostic and therapeutic challenges. However, lung functional data on COPD prevalence in CHF are scarce and COPD remains widely undiagnosed or misdiagnosed. The reported prevalence rates of COPD range from 9 to 41% in European cohorts and from 11 to 52% in North American patients with heart failure. The purpose of this study was to determine the prevalence, underdiagnosis, and overdiagnosis of COPD as determined by spirometry and according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria in patients with CHF.
3. There is abundant evidence of increased systemic inflammation in both CHF and COPD and it is remarkable to observe the similarities of inflammation in both conditions. These inflammatory responses may provide a mechanistic bridge between COPD and cardiac co-morbidity. However, there is no information regarding systemic inflammation when CHF and COPD coexist. It is unknown whether the combination of these two diseases leads to increased systemic inflammation in comparison to CHF alone. The aim of this study was to investigate the presence of systemic inflammation, as measured by inflammatory parameters (leukocytes, platelets, high sensitivity CRP), in CHF patients with or without COPD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure patients with left ventricular systolic dysfunction (left ventricular ejection fraction < 40%)
* Outpatients
* New York Heart Association (NYHA) class I-IV
* 18 years and older
* Informed consent

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Patients who are not able to cooperate or undergo pulmonary function tests
* Other diseases that can lead to obstructive lung function: asthma, cystic fibrosis
* Malignancy with bad prognosis (survival < 6 months)
* Hospitalisation to the pulmonary department in the past 6 weeks, in this case patients will have the pulmonary function tests ≥ 6 weeks after discharge
* Patients who are already participating in another study within the cardiology department

Additional exclusion criteria for the first primary objective:

* Disorders/diseases that can lead to pulmonary function impairment:

  * Pulmonary: lung surgery (lobectomy/pneumectomy), parenchymal neoplasms, interstitial lung disease, sarcoidosis, pneumoconioses, lung abscess, lobar pneumonia, post- infectious scarring, atelectasis, radiation fibrosis
  * Pleural: diffuse pleural thickening, mesothelioma, pleural effusion not due to heart failure, pneumothorax
  * Neuromuscular diseases: ALS, poliomyelitis, myopathy, bilateral diaphragmatic paralysis, high spinal cord lesions, myasthenia gravis
  * Abdominal: obesity (BMI > 35) (exclusion only from the restriction prevalence analysis)
  * Pericardial: major pericardial effusion
  * Large mediastinal processes
  * Collagen vascular diseases

Additional exclusion criteria for the third primary objective:

* Active/recent infection
* Febrile or inflammatory disease such as rheumatoid arthritis
* Use of antibiotics or anti-inflammatory medication, such as etanercept, infliximab, systemic use of corticosteroids and NSAID's other than acetylsalicylic acid
* Malignancy
* Auto-immune disease
* Collagenvascular disease
* Gastro-intestinal disease (such as inflammatory bowel disease)
* Recent operation (past 3 months)
* Renal or liver failure
* Thyroid disease
* Obstructive sleep apnoea syndrome (OSAS)
* Disorders that lead to thrombocytopenia/leukocytopenia or thrombocytosis/leukocytosis (hs-CRP analysis will take place in case these disorders do not affect hs-CRP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary function abnormalities | 1 day
  Restriction, obstruction, diffusion impairment, mixed pulmonary defects
COPD prevalence, underdiagnosis, and overdiagnosis | 3 months
  Patients with newly diagnosed COPD repeated spirometry after 3 months of standard treatment for COPD to confirm persistent airway obstruction (COPD) and thus exclude asthma.
Systemic inflammation | 1 day
  Leukocytes, platelets, high sensitivity CRP.

SECONDARY OUTCOMES:
Quality of life | 3 months
  Minnesota Living with Heart Failure Questionnaire (MLHFQ), on the day of initial pulmonary function tests and 3 months later.
Dyspnoea | 3 months
  modified Medical Research Council (MRC) dyspnea scale and 10-point Borg dyspnoea score, on the day of initial pulmonary function tests and 3 months later.
Independent predictors of COPD | 3 months
  Patients characterisitcs, such as age, gender, body mass index, symptoms, smoking history, family history, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Armine G Minasian, MD, Principal Investigator — Rijnstate Hospital, Arnhem, The Netherlands
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Rijnstate Hospital, Zevenaar, Gelderland

REFERENCES:
- [Derived] Minasian AG, van den Elshout FJ, Dekhuijzen PN, Vos PJ, Willems FF, van den Bergh PJ, Heijdra YF. Using the Lower Limit of Normal Instead of the Conventional Cutoff Values to Define Predictors of Pulmonary Function Impairment in Subjects With Chronic Heart Failure. Respir Care. 2016 Feb;61(2):173-83. doi: 10.4187/respcare.04101. Epub 2015 Oct 20. PMID 26487748
- [Derived] Minasian AG, van den Elshout FJ, Dekhuijzen PR, Vos PJ, Willems FF, van den Bergh PJ, Heijdra YF. Serial pulmonary function tests to diagnose COPD in chronic heart failure. Transl Respir Med. 2014 Dec;2(1):12. doi: 10.1186/s40247-014-0012-5. Epub 2014 Sep 25. PMID 25285269